CLINICAL TRIAL: NCT07377032
Title: L-serine Supplementation in Patients With GRIN-related Neurodevelopmental Disorders: Multicentre Protocol for an Aggregated Series of Randomised, Placebo-controlled N-of-1 Trials
Brief Title: TAP-GRIN: Interventional Study on Patients With GRIN-related Neurodevelopmental Disorders
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Meyer Children's Hospital IRCCS (Other)
Responsible Party: Principal Investigator, Simona Balestrini, MD, Meyer Children's Hospital IRCCS
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: TAP-GRIN
Record Dates: First submitted 2026-01-19; First posted 2026-01-29 (Actual); Last update posted 2026-01-29 (Actual); Status verified 2026-01

CONDITIONS: GRIN-related Disorders; GRIN1; GRIN2A; GRIN2B; GRIN2D; Epilepsy; Neurodevelopmental Disorder (Diagnosis)
MeSH Terms: conditions — Epilepsy; Neurodevelopmental Disorders; Disease | interventions — Serine; maltodextrin

STUDY DESIGN:
Intervention Model Description: Aggregated series of n-of-1 trials
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental group (Active Comparator): L-serine supplementation is administered as an oral powder for solution and used as an add-on intervention to participants' existing standard of care. L-serine is a naturally occurring amino acid and is classified as a food for special medical purposes. In this study, L-serine is used to increase the availability of its enantiomer D-serine, an endogenous co-agonist of the N-methyl-D-aspartate receptor (NMDAR), with the aim of enhancing NMDAR-mediated neurotransmission in individuals with GRIN-related neurodevelopmental disorders caused by loss-of-function variants.
  The intervention is delivered using a randomised, double-blind, placebo-controlled n-of-1 design, in which each participant receives both L-serine and placebo in alternating treatment periods. L-serine and placebo are identical in appearance, packaging, and method of administration to maintain blinding. Treatment allocation within each cycle is determined by a computer-generated randomisation schedule managed by unblinded
  Interventions: Dietary Supplement: L-serine
- Placebo (Placebo Comparator): Placebo is administered as an oral powder for solution and serves as the comparator to L-serine supplementation. The placebo consists primarily of maltodextrin, a readily digestible carbohydrate that is commonly used as an inert control substance in clinical studies. It is classified as a food-grade product and contains no active amino acids or pharmacologically active ingredients.
  The placebo is formulated to be indistinguishable from L-serine with respect to appearance, texture, solubility, and method of administration, in order to maintain blinding of participants, caregivers, investigators, and study staff. Packaging, labelling, and dosing instructions are identical to those used for the active intervention.
  The placebo is administered orally in three divided daily doses, following the same dosing schedule and duration as the active intervention within the randomised, double-blind, n-of-1 trial design. Each placebo treatment period lasts three months, with the first seven days d
  Interventions: Other: Maltodextrin (Placebo)

INTERVENTIONS:
Dietary Supplement: L-serine — L-serine supplementation is administered as an oral powder for solution and used as an add-on intervention to participants' existing standard of care. L-serine is a naturally occurring amino acid and is classified as a food for special medical purposes. In this study, L-serine is used to increase the availability of its enantiomer D-serine, an endogenous co-agonist of the N-methyl-D-aspartate receptor (NMDAR), with the aim of enhancing NMDAR-mediated neurotransmission in individuals with GRIN-related neurodevelopmental disorders caused by loss-of-function variants.
  The intervention is delivered using a randomised, double-blind, placebo-controlled n-of-1 design, in which each participant receives both L-serine and placebo in alternating treatment periods. L-serine and placebo are identical in appearance, packaging, and method of administration to maintain blinding. Treatment allocation within each cycle is determined by a computer-generated randomisation schedule managed by unblinded s
  Arms: Experimental group
Other: Maltodextrin (Placebo) — Placebo is administered as an oral powder for solution and serves as the comparator to L-serine supplementation. The placebo consists primarily of maltodextrin, a readily digestible carbohydrate that is commonly used as an inert control substance in clinical studies. It is classified as a food-grade product and contains no active amino acids or pharmacologically active ingredients.
  The placebo is formulated to be indistinguishable from L-serine with respect to appearance, texture, solubility, and method of administration, in order to maintain blinding of participants, caregivers, investigators, and study staff. Packaging, labelling, and dosing instructions are identical to those used for the active intervention.
  The placebo is administered orally in three divided daily doses, following the same dosing schedule and duration as the active intervention within the randomised, double-blind, n-of-1 trial design. Each placebo treatment period lasts three months, with the first seven days de
  Arms: Placebo

SUMMARY:
The goal of this clinical study is to find out whether L-serine dietary supplementation helps improve overall clinical functioning in children and young adults (2-30 years) with GRIN-related neurodevelopmental disorders (GRIN-NDD) caused by loss-of-function (LoF) variants in GRIN1, GRIN2A, GRIN2B, or GRIN2D. It will also assess the safety and tolerability of L-serine.

The main questions it aims to answer are:

Does L-serine improve overall clinical status, measured mainly by the Clinical Global Impression-Severity (CGI-S) score?

Does L-serine improve behaviour, cognition, adaptive functioning, motor skills, sleep, and (in those with epilepsy) seizure frequency and EEG findings?

What side effects or medical problems occur during L-serine compared with placebo?

Do neurophysiological measures (including TMS-EMG/TMS-EEG) change with treatment and potentially act as biomarkers of response?

Researchers will compare L-serine to a placebo (maltodextrin powder with similar appearance/texture) using a randomised, double-blind, placebo-controlled "n-of-1" approach, where each participant receives both treatments in alternating periods. Results from multiple single-patient trials will then be combined (aggregated) to estimate the overall treatment effect across the study population.

Participants will:

Complete a 4-week baseline period with assessments (and seizure diary use where applicable)

Receive L-serine and placebo in alternating 3-month periods within each cycle (minimum 2 cycles, up to 4 cycles; each cycle lasts 6 months)

Take the assigned study product by mouth 3 times per day at 500 mg/kg/day (maximum 30 g/day for participants ≥60 kg)

Have the first 7 days of each 3-month period treated as washout, with data from that week not analysed

Attend regular clinic visits for clinical exams, safety labs, and standardized assessments of global status, behaviour/cognition, motor function, and sleep

If they have epilepsy: keep a seizure diary and undergo EEG assessments after each treatment period

In some sites (Italy and France): undergo TMS-based neurophysiology testing

Optionally, a subset may join a cellular biomarker substudy (blood collection to generate iPSC-derived neuronal models and organoids) to explore treatment effects in variant-specific lab models.

DETAILED DESCRIPTION:
GRIN-related neurodevelopmental disorders (GRIN-NDD) are rare genetic conditions caused by pathogenic variants in GRIN1, GRIN2A, GRIN2B, or GRIN2D, which encode subunits of the N-methyl-D-aspartate receptor (NMDAR). NMDARs play a central role in synaptic transmission, plasticity, and neurodevelopment. Variants affecting these genes may result in altered receptor function, most commonly loss of function (LoF), leading to a spectrum of neurodevelopmental phenotypes that include epilepsy, intellectual disability, behavioural abnormalities, sleep disturbances, and motor impairment.

Preclinical and clinical evidence suggests that enhancement of NMDAR co-agonist availability may partially restore receptor function in individuals with LoF GRIN variants. L-serine, a naturally occurring amino acid, serves as a metabolic precursor of D-serine, a major endogenous NMDAR co-agonist. Oral L-serine supplementation has been associated with clinical improvement in small case series and early-phase clinical studies involving individuals with GRIN-NDD due to LoF variants. However, systematic evidence from randomised, blinded studies remains limited, particularly given the rarity and phenotypic heterogeneity of these disorders.

This study is designed to evaluate the clinical effect and safety of L-serine supplementation using an aggregated series of randomised, double-blind, placebo-controlled n-of-1 trials. The n-of-1 approach allows each participant to serve as their own control and is well suited to rare diseases with substantial inter-individual variability. By aggregating data from multiple single-patient trials using Bayesian hierarchical models, the study aims to provide both individual-level and population-level estimates of treatment effect.

Following a baseline observation period, participants will undergo repeated treatment cycles in which L-serine supplementation and placebo are administered in alternating periods. Each cycle consists of two treatment periods of equal duration, with the order of treatments randomised for each cycle. A short washout interval is incorporated at the start of each treatment period to minimise potential carry-over effects. Both participants and investigators remain blinded to treatment allocation throughout the study, except in cases of emergency unblinding for safety reasons.

L-serine and placebo are provided as oral powders for solution and are administered at a fixed weight-based dose divided into three daily administrations. No dose titration is planned. Concomitant treatments, including antiseizure medications and other standard therapies, are permitted and remain stable whenever clinically feasible. Participants are monitored longitudinally through scheduled visits that include clinical evaluations, safety laboratory testing, and protocol-specified assessments.

The primary focus of the study is the assessment of global clinical change associated with L-serine supplementation compared with placebo. Secondary evaluations examine treatment effects across multiple functional domains, including behaviour, cognition, adaptive functioning, motor abilities, sleep quality, and, in participants with epilepsy, seizure frequency and electroencephalographic (EEG) features. These assessments are conducted repeatedly at the end of each treatment period, enabling within-subject comparisons across treatment conditions.

In addition to clinical outcomes, the study incorporates neurophysiological assessments to explore objective biomarkers of treatment response. Transcranial magnetic stimulation (TMS) combined with electromyography (EMG) and electroencephalography (EEG) is used at selected sites to characterise cortical excitability, inhibitory and excitatory balance, and network-level responses to stimulation. These measures are intended to provide mechanistic insights into NMDAR-related cortical function and to identify potential biomarkers that correlate with clinical response to L-serine.

An optional preclinical biomarker substudy is included for a subset of participants who provide additional consent. In this substudy, peripheral blood samples are used to generate induced pluripotent stem cells (iPSCs), which are subsequently differentiated into neuronal cell models and, in selected cases, three-dimensional brain organoids. These patient-derived models are used to examine neuronal development, synaptic function, network activity, and plasticity in vitro, and to assess the effects of L-serine exposure at the cellular and molecular levels. Data from this substudy are exploratory and are intended to support translational interpretation of clinical findings.

Safety monitoring is conducted throughout the study in accordance with Good Clinical Practice principles. Adverse events are systematically collected and evaluated for severity and potential relationship to the study product. Predefined criteria are in place for treatment discontinuation and early withdrawal in the event of clinical worsening or safety concerns. Given the non-pharmacological classification of L-serine as a food for special medical purposes and its prior clinical use, no specific toxicity signals are anticipated; however, ongoing monitoring is implemented to ensure participant safety.

The study is conducted across multiple international centres with expertise in GRIN-NDD. The innovative design of aggregated n-of-1 trials is intended to maximise the interpretability of results in a rare disease context, allowing identification of both average treatment effects and inter-individual variability in response. The findings are expected to inform clinical decision-making, contribute to evidence-based use of L-serine in GRIN-NDD, and support the broader application of n-of-1 trial methodologies in rare neurological disorders.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of a GRIN-related neurodevelopmental disorder (GRIN-NDD)
* Presence of a pathogenic or likely pathogenic loss-of-function (LoF) variant in GRIN1, GRIN2A, GRIN2B, or GRIN2D
* Parent(s), caregiver(s), or legally authorised representative(s) have been informed of the nature of the study and have provided written informed consent.
* Participants who are able to do so have provided written informed consent or assent, according to local regulations and cognitive capacity.
* Parent(s)/caregiver(s) are willing and able to comply with study procedures and visits, in the opinion of the investigator.
* Participants who have previously received L-serine supplementation are willing to discontinue L-serine for at least one week prior to the baseline observation period.

Exclusion Criteria:

* Age younger than 2 years at screening.
* Known hypersensitivity or intolerance to L-serine, placebo, or any excipients used in the study formulations.
* Presence of a clinically significant unstable medical condition (other than epilepsy) that, in the investigator's judgement, may place the participant at increased risk or interfere with study participation.
* Any other significant disease or disorder that may compromise participant safety, affect study outcomes, or impair the participant's ability to complete the study procedures.
* Inadequate supervision by parent(s) or caregiver(s), as judged by the investigator.
* Participation in another clinical trial involving an investigational medicinal product within the previous 6 months.
* Female participants who are pregnant or breastfeeding.
* Presence of a GRIN1, GRIN2A, GRIN2B, or GRIN2D variant for which a clear loss-of-function effect cannot be demonstrated.

Ages: 2 Years to 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-08-29 (Actual); Primary Completion 2028-06 (Estimated); Study Completion 2028-06 (Estimated)

PRIMARY OUTCOMES:
Change in Clinical Global Impression - Severity (CGI-S) score | From baseline to the end of each 3-month treatment period, assessed repeatedly across all completed treatment cycles (minimum 2 cycles, up to 4 cycles; total study duration up to approximately 104 weeks).
  The Clinical Global Impression - Severity (CGI-S) scale is a clinician-rated measure of overall illness severity. The primary outcome is the within-subject difference in CGI-S score comparing L-serine supplementation with placebo, assessed at the end of each treatment period relative to baseline. Lower CGI-S scores indicate less severe overall clinical status.

SECONDARY OUTCOMES:
Number of adverse events | From baseline through the end of the last treatment period and the 2-week post-treatment safety follow-up (up to approximately 110 weeks).
  Safety and tolerability will be assessed through the collection of adverse events (AEs), serious adverse events (SAEs), clinical examinations, vital signs, body weight, neurological examinations, and laboratory parameters during L-serine and placebo periods.
Change in Clinical Global Impression - Improvement (CGI-I) score | Assessed at the end of each 3-month treatment period across all completed treatment cycles (minimum 2 cycles, up to 4 cycles; up to approximately 104 weeks)
  The CGI-I is a clinician-rated measure of overall improvement or worsening compared with baseline. Changes in CGI-I scores will be compared between L-serine and placebo treatment periods within subjects.
Change in behavioural functioning | From baseline to the end of each 3-month treatment period across all completed treatment cycles (up to approximately 104 weeks).
  Behavioural changes will be assessed using age-appropriate standardized instruments (Child Behavior Checklist [CBCL] or Adult Behavior Checklist [ABCL]). Scores obtained at the end of each treatment period will be compared with baseline and between L-serine and placebo periods.
Change in adaptive functioning | From baseline to the end of each 3-month treatment period across all completed treatment cycles (up to approximately 104 weeks).
  Adaptive functioning will be assessed using standardized measures (Vineland Adaptive Behavior Scales [VABS] or Adaptive Behaviour Assessment System, Third Edition [ABAS-3], as appropriate). Changes from baseline will be compared between treatment conditions.
Change in cognitive performance | From baseline to the end of each 3-month treatment period across all completed treatment cycles (up to approximately 104 weeks).
  Cognitive performance will be evaluated using EpiTrack Junior or EpiTrack, depending on participant age. Changes in total and subscale scores will be compared between L-serine and placebo treatment periods.
Change in motor function | From baseline to the end of each 3-month treatment period across all completed treatment cycles (up to approximately 104 weeks).
  Motor function will be assessed using the Manual Ability Classification System (MACS) and, when feasible, the Movement Assessment Battery for Children - Second Edition (MABC-2). Changes from baseline will be compared across treatment periods.
Change in sleep quality | From baseline to the end of each 3-month treatment period across all completed treatment cycles (up to approximately 104 weeks).
  Sleep quality will be assessed using standardized questionnaires (Pittsburgh Sleep Quality Index [PSQI] and/or age-appropriate sleep questionnaires). Changes from baseline will be compared between L-serine and placebo periods
Change in seizure frequency (epilepsy subgroup) | From baseline to the end of each 3-month treatment period across all completed treatment cycles (up to approximately 104 weeks).
  For participants with epilepsy, seizure frequency will be assessed using caregiver-completed seizure diaries. Percentage change in seizure frequency per 28 days will be compared between L-serine and placebo treatment periods.
Change in epileptiform discharge frequency on EEG (epilepsy subgroup) | From baseline to the end of each 3-month treatment period across all completed treatment cycles (up to approximately 104 weeks).
  Standard EEG recordings will be evaluated by expert review using a participant-specific scoring system (worsened, unchanged, or improved). EEG changes will be compared between L-serine and placebo periods.
Change in neurophysiological biomarkers (TMS-EMG / TMS-EEG) | From baseline to the end of each 3-month treatment period across all completed treatment cycles (up to approximately 104 weeks).
  Neurophysiological measures derived from transcranial magnetic stimulation combined with EMG and EEG will be analysed to assess changes in cortical excitability, inhibition/facilitation balance, and network-level responses.

CONTACTS AND LOCATIONS:
Locations (3):
- Hospices Civils de Lyon, Lyon, France
- Meyer Children's Hospital, Florence, Italy
- Children's Memorial Health Institute, Warsaw, Poland

IPD SHARING:
Plan to Share IPD: No